CLINICAL TRIAL: NCT06096896
Title: The Efficacy and Safety of EOB-MRI Guided Microwave Ablation for Early HCC: A Multicenter, Prospective, Observational Study
Status: Active, not recruiting | Type: Observational
Sponsor: Shandong Provincial Hospital (Other Government)
Responsible Party: Principal Investigator, Chengli Li, Director of imaging magnetic resonance interventional diagnosis and Treatment Department, Shandong Provincial Hospital, Shandong Provincial Hospital
Other Study IDs: SWYX NO 2023-1035
Record Dates: First submitted 2023-10-17; First posted 2023-10-24 (Actual); Last update posted 2023-10-24 (Actual); Status verified 2023-10

CONDITIONS: Early Hepatocellular Carcinoma
Keywords: early HCC; microwave ablation; efficacy; safety
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- single-group with MWA: 334 patients with confirmed or suspected eHCC as indicated by EOB-MRI were to be included in this study in a population with high or extremely high-risk of hepatocellular carcinoma in chronic liver disease. Then Microwave ablation (MWA) was performed under EOB-MRI guidance in patients with confirmed or suspected eHCC.
  Interventions: Procedure: MWA

INTERVENTIONS:
Procedure: MWA — Microwave ablation (MWA) was performed under EOB-MRI guidance in patients with confirmed or suspected eHCC.

SUMMARY:
HCC is one of most common causes of cancer-related death in the world due to lately diagnosis by typical hallmarks which rely on completed arterialization. So it is important to earlier diagnose and treat hypovascular early HCC(eHCC). The aim of this study is to evaluate the efficacy and safety of microwave ablation for early HCC, also to explore the feasibility of EOB-MRI (Gd-EOB-DTPA enhanced MRI) guided ablation.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years;
2. Patients with chronic liver disease who are at high/extremely high-risk of hepatocellular carcinoma;
3. EOB-MRI suggestive of confirmed or suspected eHCC (single lesion ≤ 2 cm or number of lesions ≤ 3 and maximum diameter ≤ 2 cm)
4. No previous history of hepatocellular carcinoma;
5. Not receiving any anti-cancer treatment;
6. Liver function Child-push A or B.

Exclusion Criteria:

1. Presence of lymph nodes or distant metastases;
2. Presence of liver metastases;
3. Prior malignancy;
4. Severe cardiopulmonary or renal dysfunction;
5. Suffering from uncorrectable coagulation dysfunction (prothrombin time > 25 seconds, prothrombin activity < 40%, platelet count ≤ 50x10^9/L);
6. Severe infectious lesions in the area of the puncture needle tract.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic liver disease at high-risk or extremely high-risk of hepatocellular carcinoma and EOB-MRI shows a confirmed or suspected eHCC.
Sampling Method: Non-Probability Sample
Enrollment: 334 (Estimated)
Dates: Start 2023-08-30 (Actual); Primary Completion 2025-09-30 (Estimated); Study Completion 2030-09-30 (Estimated)

PRIMARY OUTCOMES:
5-years overall survival (OS) after MWA for early HCC | 5 years
  Analyze the efficacy and safety of EOB-MRI-guided microwave ablation in the treatment of eHCC;

SECONDARY OUTCOMES:
Rate of completed ablation after MWA | rate of completed ablation at one month
  Ablation effect assessed by EOB-MRI one month after ablation

CONTACTS AND LOCATIONS:
Locations (1):
- Shandong PH, Jinan, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Llovet JM, Kelley RK, Villanueva A, Singal AG, Pikarsky E, Roayaie S, Lencioni R, Koike K, Zucman-Rossi J, Finn RS. Hepatocellular carcinoma. Nat Rev Dis Primers. 2021 Jan 21;7(1):6. doi: 10.1038/s41572-020-00240-3. PMID 33479224
- [Result] International Consensus Group for Hepatocellular NeoplasiaThe International Consensus Group for Hepatocellular Neoplasia. Pathologic diagnosis of early hepatocellular carcinoma: a report of the international consensus group for hepatocellular neoplasia. Hepatology. 2009 Feb;49(2):658-64. doi: 10.1002/hep.22709. No abstract available. PMID 19177576
- [Result] Sirlin CB, Kielar AZ, Tang A, Bashir MR. LI-RADS: a glimpse into the future. Abdom Radiol (NY). 2018 Jan;43(1):231-236. doi: 10.1007/s00261-017-1448-1. PMID 29318354
- [Result] Omata M, Cheng AL, Kokudo N, Kudo M, Lee JM, Jia J, Tateishi R, Han KH, Chawla YK, Shiina S, Jafri W, Payawal DA, Ohki T, Ogasawara S, Chen PJ, Lesmana CRA, Lesmana LA, Gani RA, Obi S, Dokmeci AK, Sarin SK. Asia-Pacific clinical practice guidelines on the management of hepatocellular carcinoma: a 2017 update. Hepatol Int. 2017 Jul;11(4):317-370. doi: 10.1007/s12072-017-9799-9. Epub 2017 Jun 15. PMID 28620797
- [Result] Choi JY, Lee JM, Sirlin CB. CT and MR imaging diagnosis and staging of hepatocellular carcinoma: part I. Development, growth, and spread: key pathologic and imaging aspects. Radiology. 2014 Sep;272(3):635-54. doi: 10.1148/radiol.14132361. PMID 25153274
- [Result] Renzulli M, Biselli M, Brocchi S, Granito A, Vasuri F, Tovoli F, Sessagesimi E, Piscaglia F, D'Errico A, Bolondi L, Golfieri R. New hallmark of hepatocellular carcinoma, early hepatocellular carcinoma and high-grade dysplastic nodules on Gd-EOB-DTPA MRI in patients with cirrhosis: a new diagnostic algorithm. Gut. 2018 Sep;67(9):1674-1682. doi: 10.1136/gutjnl-2017-315384. Epub 2018 Feb 3. PMID 29437912
- [Result] Reig M, Forner A, Rimola J, Ferrer-Fabrega J, Burrel M, Garcia-Criado A, Kelley RK, Galle PR, Mazzaferro V, Salem R, Sangro B, Singal AG, Vogel A, Fuster J, Ayuso C, Bruix J. BCLC strategy for prognosis prediction and treatment recommendation: The 2022 update. J Hepatol. 2022 Mar;76(3):681-693. doi: 10.1016/j.jhep.2021.11.018. Epub 2021 Nov 19. PMID 34801630
- [Result] Kudo M, Kawamura Y, Hasegawa K, Tateishi R, Kariyama K, Shiina S, Toyoda H, Imai Y, Hiraoka A, Ikeda M, Izumi N, Moriguchi M, Ogasawara S, Minami Y, Ueshima K, Murakami T, Miyayama S, Nakashima O, Yano H, Sakamoto M, Hatano E, Shimada M, Kokudo N, Mochida S, Takehara T. Management of Hepatocellular Carcinoma in Japan: JSH Consensus Statements and Recommendations 2021 Update. Liver Cancer. 2021 Jun;10(3):181-223. doi: 10.1159/000514174. Epub 2021 May 19. PMID 34239808
- [Result] Facciorusso A, Abd El Aziz MA, Tartaglia N, Ramai D, Mohan BP, Cotsoglou C, Pusceddu S, Giacomelli L, Ambrosi A, Sacco R. Microwave Ablation Versus Radiofrequency Ablation for Treatment of Hepatocellular Carcinoma: A Meta-Analysis of Randomized Controlled Trials. Cancers (Basel). 2020 Dec 16;12(12):3796. doi: 10.3390/cancers12123796. PMID 33339274
- [Result] Chen L, Ren Y, Sun T, Cao Y, Yan L, Zhang W, Ouyang T, Zheng C. The efficacy of radiofrequency ablation versus cryoablation in the treatment of single hepatocellular carcinoma: A population-based study. Cancer Med. 2021 Jun;10(11):3715-3725. doi: 10.1002/cam4.3923. Epub 2021 May 7. PMID 33960697
- [Result] Suwa K, Seki T, Aoi K, Yamashina M, Murata M, Yamashiki N, Nishio A, Shimatani M, Naganuma M. Efficacy of microwave ablation versus radiofrequency ablation for hepatocellular carcinoma: a propensity score analysis. Abdom Radiol (NY). 2021 Aug;46(8):3790-3797. doi: 10.1007/s00261-021-03008-9. Epub 2021 Mar 6. PMID 33675382
- [Result] Wang F, Numata K, Nihonmatsu H, Chuma M, Moriya S, Nozaki A, Ogushi K, Fukuda H, Ruan L, Okada M, Luo W, Koizumi N, Nakano M, Otani M, Inayama Y, Maeda S. Intraprocedurally EOB-MRI/US fusion imaging focusing on hepatobiliary phase findings can help to reduce the recurrence of hepatocellular carcinoma after radiofrequency ablation. Int J Hyperthermia. 2020;37(1):1149-1158. doi: 10.1080/02656736.2020.1825837. PMID 32996799